CLINICAL TRIAL: NCT03586219
Title: Evaluating the Effect of Preoperative Patient Education on Postoperative Opioid Consumption, Storage, and Disposal After Urogynecologic Procedures
Brief Title: Postoperative Opioid Consumption After Urogyneocologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-4003
Record Dates: First submitted 2018-03-12; First posted 2018-07-13 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: Surgery; Patient Education; Opioid; Medication Storage; Medication Disposal
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: This is a randomized, non-blinded, controlled trial that will be performed at two sites. Study subjects will be randomized to either the control arm (standard perioperative instructions) or intervention arm (standard perioperative instructions with additional perioperative opioid-specific education) using a randomization program in a 1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Standard preoperative and postoperative instructions will be provided to the study subjects
- Intervention Arm (Experimental): Intervention: Study subjects will receive opioid-specific educational patient pamphlets in addition to standard preoperative and postoperative instructions
  Interventions: Behavioral: Opioid-specific educational patient pamphlets

INTERVENTIONS:
Behavioral: Opioid-specific educational patient pamphlets — See prior description
  Arms: Intervention Arm

SUMMARY:
The purpose of this randomized controlled trial is to evaluate whether preoperative opioid education will reduce postoperative opioid consumption after urogynecologic surgeries. Additionally, the effect of the opioid education on opioid storage and disposal patterns will be evaluated. The pattern of opioid consumption 2 and 6 weeks after surgery will be compared between patients in the study arms. The rates of prescription refills 12 weeks and 12 months after the surgery will be compared between patients in the study arms.

DETAILED DESCRIPTION:
The study concept would be introduced to the patients at the prior to or during the preoperative visit. If the patient agrees to participation during any of these encounters, written consent and HIPPA authorization will be obtained and the patient would be randomized to the intervention or control arm using a computerized randomization scheme on REDCap. The randomization will be stratified by hospital system the surgery was performed within (UC Irvine Medical Center versus Kaiser Permanente Southern California). If the patient is randomized to the intervention arm, the first opioid informational pamphlet will be provided and reviewed with the patient in addition to standard preoperative instructions. If the patient is randomized to the control arm, standard preoperative instructions will be provided. Patients within both arms of the study will receive standardized postoperative medication prescriptions prior to the surgery. Patients within both arms of the study will complete the modified surgical pain score and preoperative opioid education study survey prior to surgery.

After the surgery is completed, the primary surgeon will decide whether to admit the patient to the hospital and which postoperative analgesics will be administered within the hospital prior to discharge for subjects in both study arms. The patient will follow up for standard postoperative clinic visits at 2 weeks and 6 weeks postoperatively. One to two days prior to the 2 week postoperative visit, the patients will be contacted via telephone to remind them to bring their opioid prescription bottles to the clinic visit.

Between the surgery date and the 2 week postoperative visit, the electronic medical records will be reviewed to evaluate the length of the surgery, intraoperative complications, the postoperative date of discharge, the postoperative date of removal of the transurethral foley catheter, the total daily morphine equivalents that the patient was prescribed prior to discharge from the hospital, and the presence of opioid prescriptions 30 days prior to the surgery. Additionally, the CURES 2.0 Database will be queried to evaluate for opioid prescriptions 30 days prior to the surgery.

During the 2 week postoperative visit, the remaining opioid tablets will be counted and recorded by a co-investigator. The patient will complete the modified surgical pain score and postoperative opioid education study survey. The electronic medical record system and CURES 2.0 Database will be queried to evaluate for additional opioid prescriptions since the time of surgery. Patients randomized to the intervention arm will receive the second opioid informational pamphlet, which will be reviewed by a co-investigator.

During the 6 week the patient will complete the modified surgical pain score and postoperative opioid education study survey. The electronic medical record system and CURES 2.0 Database will be queried to evaluate for additional opioid prescriptions since the time of surgery. The patients' electronic medical records will be reviewed after the 6 week postoperative visit to evaluate for postoperative complications.

Twelve week after the surgery, the electronic medical record system and CURES 2.0 Database will be queried to evaluate for additional opioid prescriptions since the time of surgery.

If a patient fails to follow up for a postoperative visit, at least two attempts will be made to contact the patient via telephone to collect opioid pill counts and have the patient verbally complete the modified surgical pain score and postoperative opioid education study survey. Initial statistical analysis will be performed after the 12 week postoperative review of the electronic medical records and CURES 2.0 Database have been completed.

Twelve months after the surgery, the electronic medical record system and CURES 2.0 Database will be queried to evaluate for additional opioid prescriptions since the time of surgery. Additional statistical analysis will be performed after the 12 month opioid refill prescriptions have been evaluated.

While this is a multi-site trial involving subjects from UC Irvine Medical Center, Kaiser Permanente Orange County - Irvine, and Kaiser Permanente Orange County - Anaheim, only de-identified data will be uploaded into the REDCap data management system. The lead investigator will maintain a separate key containing patient health information for subjects from both sites, which will be utilized to evaluate for additional opioid prescriptions 12 months after the surgery. Co-investigators from both study sites will not have access to identifiable data from subjects that were not recruited from their particular study site.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-99 years old
* English speaking
* Evaluated by a provider within the Urogynecology division at UC Irvine Medical Center, Kaiser Permanente Orange County - Irvine Medical Center, or Kaiser Permanente Orange County - Anaheim Medical Center, and consented for either a uterosacral ligament suspension, sacrospinous ligament fixation, minimally-invasive colpopexy (either laparoscopic or robotic-assisted laparoscopic), colporrhaphy, or colpocleisis

Exclusion Criteria:

* Non English-speaking
* Cognitive deficits that would prevent the patient from completing the study questionnaires
* Cancellation of the surgery
* Combined case with another surgical service (i.e. colorectal surgery)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients who are undergoing either reconstructive or obliterative surgeries for the indication of pelvic organ prolapse. Patients who identify as female but do not have the predisposing condition of pelvic organ prolapse will not be recruited.
Enrollment: 146 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-11-28 (Actual)

PRIMARY OUTCOMES:
2 week postoperative opioid consumption | 2 weeks after the surgery
  Mean number of opioid tablets consumed 2 weeks postoperatively

SECONDARY OUTCOMES:
Modified Surgical Pain Score | Between the preoperative assessment and 6 weeks after surgery
  To be collected at the preoperative assessment and 2 weeks and 6 weeks after surgery. This is a 4 question score that evaluates pain at rest, with normal activities, with strenuous activities, and quantifies bother or discomfort associated with the pain. A numerical answer for each question is selected from a 10 point scale ranging from 0 (no pain or bother) to 10 (maximum pain or bother). Higher scores are associated with worse outcomes.
Preoperative Patient Survey answers | To be collected within 30 days prior to surgery. This data point will be included in the initial analysis that will be performed after the last enrolled patient has completed the 12 week postoperative chart review.
  Investigator-initiated survey to assess for chronic pain conditions and general understanding of opioid disposal patterns
Postoperative Patient Survey answers | Conducted two times 2 weeks and 6 weeks after surgery. This data point will be included in the initial analysis that will be performed after the last enrolled patient has completed the 12 week postoperative chart review.
  Investigator-initiated survey assessing patient satisfaction with opioid prescription, storage and disposal patterns, that will be conducted at 2 weeks, 6 weeks, and 12 weeks after the surgery
Additional opioid prescriptions | To be performed three times between 2 weeks to 12 months after the surgery. This data point will be included in the initial analysis that will be performed after the last enrolled patient has completed the 12 week postoperative chart review.
  The electronic medical records at each site, as well as the California Department of Justice CURES 2.0 database will be evaluated 2 weeks, 6 weeks, 12 weeks, and 12 months after the surgery
Intraoperative complications | These will be evaluated within the first 6 weeks after surgery. This data point will be included in the initial analysis that will be performed after the last enrolled patient has completed the 12 week postoperative chart review.
  Defined as the presence of packed red blood cell transfusion, bowel injury, bladder injury, ureteral injury, or conversion to laparotomy
Postoperative complications | The electronic medical record will be reviewed 6 weeks after surgery. This data point will be included in the initial analysis that will be performed after the last enrolled patient has completed the 12 week postoperative chart review.
  Defined as either the presence of mesh exposure, wound infection, packed red blood cell transfusion, neuropathy, or urinary tract infection within 6 weeks postoperatively or return to the operating room for within 14 days post operatively
Postoperative Oral Morphine Equivalents Prior to Discharge | The electronic medical record will be reviewed 2 weeks after surgery. This data point will be included in the initial analysis that will be performed after the last enrolled patient has completed the 12 week postoperative chart review.
  Total daily oral morphine equivalents prescribed in the hospital prior to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Buono, MD, Principal Investigator — University of California, Irvine
Locations (3):
- United States (3):
  - Kaiser Permanente Orange County - Anaheim, Anaheim, California
  - Kaiser Permanente Orange County-Irvine Medical Center, Irvine, California
  - University of California Irvine Medical Center, Orange, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buono K, Whitcomb E, Guaderrama N, Lee E, Ihara J, Sudol N, Lane F, Lee J, Heliker BD, Brueseke T. A Randomized Controlled Trial Assessing the Impact of Opioid-Specific Patient Counseling on Opioid Consumption and Disposal After Reconstructive Pelvic Surgery. Female Pelvic Med Reconstr Surg. 2021 Mar 1;27(3):151-158. doi: 10.1097/SPV.0000000000001009. PMID 33620897

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT03586219/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT03586219/ICF_001.pdf